CLINICAL TRIAL: NCT03641443
Title: Non-Invasive Measurement of Absolute Intracranial Pressure in Patients With Mass Effective Brain Tumors
Brief Title: non_invasive_aICP_Tumor
Acronym: aICPTumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Javier Fandino, MD, MD, Kantonsspital Aarau
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: aICP Tumor
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Tumor, Brain; Intracranial Pressure Increase
MeSH Terms: conditions — Brain Neoplasms; Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-invasive measurement of intracranial pressure (Experimental): Patient with mass effective brain tumor that undergo non-invasive intracranial pressure measurement
  Interventions: Device: Non-invasive measurement of intracranial pressure

INTERVENTIONS:
Device: Non-invasive measurement of intracranial pressure — Non-invasive measurement of intracranial pressure in patients with mass effective brain Tumors

SUMMARY:
Since decades, neurosurgeons and neurooncologists assumed that the mass effect of brain tumors with peritumoral edema or intratumoral hemorrhage might lead to increased ICP. Therefore, decisions on surgical procedures and medical treatments were made based on clinical and radiological findings suggesting increased ICP. But in fact, no measurement has ever confirmed increased ICP in brain tumor patients. From an ethical point of view, it is not justifiable to implant an intraparenchymal ICP probe within an invasive surgical procedure in a brain tumor patient unless the patient is comatose or present with rapid impairment of the level of consciousness. Therefore, with the new medical device for non-invasive ICP measurement presented in this study protocol, we will be able to measure absolute ICP values in patients with brain tumors.

DETAILED DESCRIPTION:
Primary brain tumors in adults are less common than metastatic tumors. The most frequent are glioblastoma multiforme, metastases, anaplastic astrocytoma, meningioma, pituitary tumors and vestibular schwannoma. 70% of the tumors in adults are supratentorial. The most infratentorial tumors are metastases, schwannoma, meningioma, epidermoid, hemangioblastoma, and brainstem glioma. Causes of brain tumors are genetics, radiation, immunosuppression, viruses and chemotherapy.

Clinically patients present with neurological deficits as hemiparesis, cranial nerve deficiency or signs of raised ICP such as headache, nausea, vomitus, vigilance disturbance. After clinical assessment, standard MRI with contrast agent is performed to visualize the size and structure of the tumor, contrast uptake, peritumoral edema (PTE), and other radiological findings. Depending on the tumor, size and location, the further procedure must be defined with either surgical resection, observation, other adjuvant therapies. Mostly, a histological diagnosis is needed to know the tumor biology and set supplementary treatment.

In patients with brain tumors with mass effect and peritumoral edema with consecutive midline shift increased intracranial pressure (ICP) is usually considered. During the expansion of an intracranial mass lesion, there is initially a minimal increase in ICP, but as compensatory capacity is exhausted the volume pressure curve rapidly steepens, and by further expansion of the mass a distinct increase in ICP results.

Supratentorial tumors can produce significant mass effect in the brain. In certain tumor types, especially metastases, high grade gliomas, and meningeomas significant peritumoral edema that lead to elevation of intracranial pressure might be associated. In cases of infratentorial tumors with or without edema earlier clinical decompensation with hydrocephalus, increased ICP and downward herniation are more often due to reduced space within the posterior fossa. Within the closed bony cranium, increase of volume, such as tumor with associated edema or hemorrhage, ischemia, occlusion of venous perfusion or hydrocephalus lead to an increase of ICP and secondary injury to the normal brain. PTE is caused by vasogenic edema in particular, but also cytotoxic edema, tumor-related-pressure, arterial blood supply, venous congestion and secretion of angiogenic factors such as vascular endothelial growth factor (VEGF). VEGF, Aquaporin-4 (AQP4), cyclooxygenase-2 (COX- 2), and nitric oxide (NO) induce dysfunction of tight junction proteins playing an important role in the formation of edema. Cerebral edema induced by brain tumor is characterized by an increase in the permeability of brain capillary endothelial cells and an increase in the brain water content. Peritumoral vasogenic edema as a result of blood-brain-barrier dysfunction within the tumor affects neurological function and quality of life, and may even cause life-threatening raised intracranial pressure.

Cerebral blood flow (CBF) and the carbon dioxide (CO2) reactivity, are known to be reduced in patients with brain tumor, especially those with pronounced signs of intracranial hypertension.The study reported by Chang et al. showed, that the mean CBF of both hemispheres in each group was not significantly different from brain tumor patients with peritumoral edema to age-matched controls. Cerebrovascular reactivity (CVR) was preserved in patients with mild peritumoral edema but was significantly reduced in patients with moderate and severe peritumoral edema. Surgical removal of the tumor significantly improved the impaired CVR, although the mean CBF did not change.

An earlier study on measurements of intratumoral and peritumoral blood flow as well as within the hemispheres indicated, very low flow values in the peritumoral edematous area. These findings suggest that the hypodense area surrounding brain tumor may actually represent tumor pressure ischemia.

Certain risk factors for increased edema, such as age, sex, tumor size, neurological symptoms, seizures, location, histology, and contrast enhancement, have been identified. The extend of PTE has been demonstrated as a predictor of favorable overall survival time in patients with larger PTE in metastases, but on the contrary smaller PTE was a statistically significant predictor of longer survival in high-grade gliomas. On the other hand it has been shown, that postoperative complications were more frequent and duration of intensive care treatment was longer in patients with PTE. Outcome was significantly better in patients without PTE.

Steroids are in use since 1960's and play a substantial role in the management of brain tumor and increased ICP associated with perilesional edema. Vasogenic edema responds very well to corticosteroids, although they have important side effects. Corticosteroids should be used in a low dose daily to avoid serious side effects such as myopathy, diabetes, hypertonia, osteoporosis, psychiatric alterations, skin thinning and an increased risk for some opportunistic infections.

In the study of Skjoeth et al., brain tumor patients with a substantial amount of edema were included. The effect of steroids was monitored during 5 days by clinical examination and epidural ICP measurement. ICP reduction was found only in 4 of 13 patients, another 4 patients with meningioma had a significant increase of ICP and none of them experienced clinical improvement.

Cerebral swelling through the craniotomy can seriously threaten surgical access and increase the risk of cerebral ischemia with potential worsening of outcome. Rasmussen et al. observed that subdural ICP is the strongest predictor of intraoperative brain swelling. In addition midline shift, diagnosis of glioblastoma multiforme and metastasis were significant risk factors of intraoperative brain swelling. With an intraoperative ICP greater than 13 mmHg, supra- and infratentorial brain swelling occurred with 95% probability and at an ICP greater than 26 mmHg, severe brain swelling occurred with 95% probability.

Cold et al. reported subdural ICP measurements in 29 patients during supra- and infratentorial craniotomies. The authors observed, that at subdural ICP < 6 mmHg intraoperative brain herniation never occurred. Patients with a subdural ICP greater than 7 mmHg some brain herniation was documented in all cases, and if subdural ICP was greater than 11 mmHg, pronounced brain swelling/herniation occurred in all patients. In a follow-up study, including patients receiving supratentorial craniotomy cerebral herniation did not occur at subdural ICP < 7 mmHg. On the other hand, at ICP >10 mmHg cerebral herniation occurred with high probability. These thresholds were independent of anesthetic agent used and the level of partial pressure of carbon dioxide (PCO2). Jorgensen et al. reported results of posterior fossa craniotomies where at an ICP < 10 mmHg, brain swelling/herniation rarely occurred, while at ICP ≥10 mmHg some degree of brain swelling/herniation was always present. Interestingly neurosurgeons' tactile estimation of dural tension correlated poorly with any tendency to brain swelling/herniation.

Peritumoral edema is considered to decrease after surgical resection, but there are cases where the edema enlarges postoperatively. Ono and other authors presented cases with postoperative progressive edema. Correlating to this results, it has been proven, that postoperative sustained ICP elevation occurs and the rise in ICP occurred before any neurological deterioration was noticed. Similarly, studies showed, that edema increases after radiotherapy or radiosurgery.

Although it is suspected that intracranial lesion with mass effect might cause increased ICP, there is no clinical evidence proven yet. Raised ICP can cause clinical manifestations and symptoms such as headache, nausea, vomiting, and neurological deficits. These signs, which are known as intracranial hypertension signs, are variable and have not been validated due to the lack of technological tools to measure ICP non-invasively. To date, only intra- and postoperative measurements of increased ICP have been shown with intraparenchymal ICP probes or intraventricular catheters.

The inspection of the ocular fundus would be an option to detect papilledema as a sign of intracranial hypertension. Nevertheless, papilledema is considered to have a late onset since it takes some time to be developed and not all patients with brain tumors present with fundus abnormalities. Moreover, if the patient has a preexisting condition such as high blood pressure causing intracranial hypertension and chronic papilledema, it will be difficult to assess the changes.

Currently, ICP can be measured and registered only using invasive techniques. The two ICP measurement methods available - intraventricular and intraparenchymal - require both a neurosurgical procedure, in order to implant the catheter and probes within the brain parenchyma and ventricles. Thus, these measures include themselves a risk for the subject. Infections and intracranial bleedings related to invasive ICP measurement techniques are considered frequent complications. In addition, invasive recording of ICP requires neurosurgical expertise and intensive care unit (ICU) facilities. Present review articles conclude that there is still a lack of non-invasive techniques for accurate measurement of the ICP.

Intracranial pressure (ICP) measurement is clinically important in several pathophysiology conditions. Cerebrospinal fluid (CSF) pressure is the reference for the "gold standard" invasive ICP measured via a brain ventriculostomy or by lumbar puncture in patients with free CSF circulation. Elevated ICP is a critical indication for treatment of patients with acute neurologic condition, and the best approach to management is considered to be different depending on the underlying pathophysiology. ICP can only be measured using invasive methods in routine clinical practice. The most common application of ICP monitoring is in the management of patients with severe closed head injury or some other neurologic disorders.

The concept of non-invasive ICP measurement has been discussed since the 1980s. Numerous methods for finding the objects or physiological characteristics of cerebrospinal system that would be related to the ICP and its monitoring have been postulated by many authors. Most of the proposed technologies were based on ultrasound and were capable of monitoring blood flow in intracranial or intraocular vessels, cranium diameter, or acoustic properties of the cranium. Broad research has extended into sonography of optic nerve sheath and its relation with elevated ICP. However, most of these correlation-based methods had the same problem - the need of individual patient specific calibration.

Seeking to measure absolute ICP values, researchers from Kaunas University of Technology created a non-invasive method, which does not need a patient specific calibration. The method is based on direct comparison of ICP value with the value of pressure Pe that is externally applied to the tissues surrounding the eyeball. Intracranial segment of ophthalmic artery (OA) is used as a natural sensor of ICP and extracranial segment of OA is used as a sensor of Pe. A special two depth transcranial Doppler (TCD) device is used as a pressure balance indicator when ICP = Pe. Accuracy, precision, sensitivity, specificity, and diagnostic value of this method were proven with patients with mild neurological diseases. This device has not yet been used in clinical studies to investigate ICP in brain tumor patients. A study of our neurosurgical department to validate the accuracy of non-invasive ICP measurement compared to invasive measurement techniques is ongoing.

Since decades, neurosurgeons and neurooncologists assumed, that the mass effect of brain tumors with peritumoral edema or intratumoral hemorrhage might lead to increased ICP. Therefore, decisions on surgical procedures and medical treatments were made based on clinical and radiological findings suggesting increased ICP. But in fact, no measurement has ever confirmed increased ICP in brain tumor patients. From an ethical point of view, it is not justifiable to implant an intraparenchymal ICP probe within an invasive surgical procedure in a brain tumor patient unless the patient is comatose or present with rapid impairment of the level of consciousness. Therefore, with the new medical device presented in this study protocol, we will be able to measure absolute ICP values in patients with brain tumors. The aim of the study is to correlate absolute ICP values with clinical and radiological (tumor size, midline shift and peritumoral edema) parameters which are defined as intracranial hypertension signs in brain tumor patients. The observations obtained in this study have important clinical implications to neurosurgeons, neurologists, and neurooncologists in order to define the timing of surgical procedures, medical treatments such as steroids and osmotic agents and indications for monitoring in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosed brain tumor with signs of mass effect, occlusive hydrocephalus, and/or perilesional brain edema on CT scan or magnetic resonance imaging (MRI).
* Clinical symptoms for intracranial hypertension such as headache, nausea, vomiting, neurological deficits, cognitive deficits, hemiparesis or cranial nerve deficits.
* Age: ≥ 18 years at admission
* Informed consent

Exclusion Criteria:

* Patients with wounds, scars including the front orbital region.
* Patients with any known ocular condition that may be worsened by sustained eye pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
non-invasive, absolute intracranial pressure (aICP) before brain tumor surgery | 3 Years
  The primary outcome is the non-invasive, absolute intracranial pressure (aICP) before brain tumor surgery, as determined by the "NON-INVASIVE ICP ABSOLUTE VALUE METER" in mmHG.

SECONDARY OUTCOMES:
Correlation between increased aICP and clinical and radiological signs | 3 Years
  The secondary outcome is to demonstrate correlation between increased aICP and clinical and radiological signs.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Kienzler, MD, Principal Investigator — Kantonsspital Aarau
Locations (1):
- Kantonsspital Aarau, Aarau, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No